CLINICAL TRIAL: NCT00903292
Title: Tailored Second Line Treatment by EGFR Mutation in Patients With Advanced Lung Adenocarcinoma
Brief Title: Tailored Second Line Treatment by Epidermal Growth Factor Receptor (EGFR) Mutation in Patients With Advanced Lung Adenocarcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Wu- Chou Su, National Cheng-Kung University Hospital
Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: HR98004
Record Dates: First submitted 2009-05-15; First posted 2009-05-18 (Estimated); Last update posted 2009-05-18 (Estimated); Status verified 2009-05

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: EGFR; NSCLC; EGFR mutation rate
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A, erlotinib (Active Comparator): If EGFR mutation found then assigned to thyrosine kinase inhibitor (erlotinib)
  Interventions: Drug: erlotinib (Tarceva)
- B, pemetrexed (Active Comparator): If EGFR wild type found then assigned to chemotherapy (pemetrexed)
  Interventions: Drug: pemetrexed (Alimta)

INTERVENTIONS:
Drug: erlotinib (Tarceva) — chemotherapy with erlotinib
  Arms: A, erlotinib
Drug: pemetrexed (Alimta) — Chemotherapy with pemetrexed
  Arms: B, pemetrexed

SUMMARY:
Currently the investigators have two different classes of second-line treatment options in recurrent non-small Cell Lung Cancer (NSCLC). In chemotherapy, docetaxel and pemetrexed produced similar treatment efficacy outcomes, while pemetrexed had a better tolerability. In recent analysis of pemetrexed clinical studies, a strong treatment-by-histology interaction in overall survival and progression free survival that indicated better efficacy for non-squamous patients treated with pemetrexed. These data supports that pemetrexed could be a preferable chemotherapy drug especially in adenocarcinoma NSCLC patients.

DETAILED DESCRIPTION:
On the other hand, EGFR TKI (gefitinib or erlotinib) both produced somewhat similar higher response rate (around 25%) in general Taiwan adenocarcinoma NSCLC patients, while the median overall survival time didn't longer than chemotherapy treated patients. A recent prospective study of gefitinib in chemonaive adenocarcinoma NSCLC patients showed that the objective response rate was lower to be only 1.1% among EGFR mutation negative patients.

Since typical EGFR gene mutations (i.e., the deletion of typically five amino acids at codons 746-750 (ELREA) in exon 19 and a leucine-to-arginine mutation at codon 858 (L858R)) are a good predictor for tumor response to tyrosine kinase inhibitor, this present study is to tailor the patient's treatment according to his/her EGFR gene mutation status. Receptor tyrosine kinase inhibitor (erlotinib in this study) will be the suggested second-line drug of recommendation for typical EGFR gene mutation patients, and chemotherapy (pemetrexed in this study) will be the suggested second-line drug of recommendation for EGFR wild type patients.

The aim of this study is to increase the overall tumor response rate to 40% from current treatment outcome (around 25%) by this tailored second line treatment. The further interests of this study include prospectively evaluate the predictivity of EGFR gene mutation to tumor response.

The primary objective of this study is to determine the overall tumor response rate of tailored second line treatment determined by typical EGFR gene mutation in patients with advanced lung adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of adenocarcinoma of NSCLC.
* Locally advanced or metastatic disease (stage IIIB or IV), defined by the American Joint Committee on Cancer Staging Criteria for NSCLC (Fleming et al. 1997; Mountain 1997)
* Patients must have previously received one chemotherapy regimen for palliative therapy of locally advanced or metastatic disease.

  * NOTE: First-line therapy with a tyrosine kinase inhibitor alone or regimens including pemetrexed, docetaxel, cetuximab, and trastuzumab is not allowed for enrollment in this study.
  * Prior chemotherapy for earlier stage disease is allowed, but only a single regimen is allowed for prior palliative therapy of locally advanced or metastatic disease.
* Prior chemotherapy must be completed at least 2 weeks prior to study enrollment and the patient must have recovered from the acute toxic effects of the treatment.
* Disease status must be that of measurable disease as defined by RECIST criteria (Therasse et al. 2000).
* Performance status of 0 to 2 on the ECOG Scale (See Protocol Attachment 2.).
* Estimated life expectancy of at least 8 weeks.
* Adequate organ function including the following:

  * Bone marrow: absolute neutrophil count (ANC) 1.5* 109/L, platelets 100*109/L, hemoglobin 9 g/dL.
  * Hepatic: bilirubin 1.5ULN, AST and ALT 2.5 ULN (AST, ALT 5 ULN is acceptable if liver has tumor involvement).
  * Renal: serum creatine 1.5 ULN; Calculated creatinine clearance 45 mL/min (using the standard Cockcroft-Gault formula; Cockcroft and Gault 1976).
* For women: Must be surgically sterile, post-menopausal, or compliant with a medically approved contraceptive regimen during and for 6 months after the treatment period; must have a negative serum or urine pregnancy test and must not be lactating.
* For men: Must be surgically sterile, or compliant with a contraceptive regimen during and for 6 months after the treatment period.
* Men or women of at least 20 years of age, and signed informed consent from the patient.

Exclusion Criteria:

* Subject has untreated brain or meningeal metastases.

  * CT scans are not required to rule out brain or meningeal metastases unless there is a clinical suspicion of central nervous system disease).
  * Subjects with treated brain metastases that are radiographically or clinically stable for at least 2 weeks after therapy and have no evidence of cavitation or hemorrhage in the brain lesion are eligible providing that they are asymptomatic.
* Have previously completed or withdrawn from this study, or received pemetrexed, thymidylate synthetase or dihydrofolate reductase previously outside this study.
* Concurrent administration of any other tumor therapy.
* Active infection (at the discretion of the investigator).
* History of significant neurological or mental disorder, including seizures or dementia.
* Second primary malignancy that is clinically detectable within 5 years of consideration for study enrollment.
* Have received treatment within the last 30 days with a drug that has not received regulatory approval (e.g., warfarin or Coumadin) for any indication at the time of study entry.
* Inability to interrupt aspirin or other nonsteroidal anti-inflammatory drugs (NSAIDs) 2 days before, the day of, and 2 days after the dose of pemetrexed.

  * If a patient is taking an NSAID (Cox-2 inhibitors included) or salicylate with a long half-life (e.g., naproxen, piroxicam, diflunisal, nabumetone, rofecoxib, or celecoxib) it should not be taken 5 days before, the day of, and 2 days after the dose of pemetrexed.
* Inability or unwillingness to take erlotinib, folic acid, vitamin B12 supplementation, or dexamethasone.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-04 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
The primary analysis will be the overall best response rate, including a 95% confidence interval (Leemis and Trivedi 1996). | 02/2009 - 04/2010

CONTACTS AND LOCATIONS:
Overall Officials: Wu-Chou Su, PhD, Principal Investigator — National Cheng-Kung University Hospital
Locations (1):
- National Cheng-Kung University Hospital, Tainan, Taiwan